CLINICAL TRIAL: NCT03672825
Title: RECLAIM: A Phase I Safety and Feasibility Trial of REcycled CartiLage Auto/Allo IMplantation for the Treatment and Repair of Focal Knee Cartilage Defects
Brief Title: REcycled CartiLage Auto/Allo IMplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aaron Krych, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-000939
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Cartilage Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RECLAIM (Experimental): Treating cartilage defects with autologous (your own) cartilage cells mixed with allogeneic (from someone else) adipose-derived mesenchymal stem cells (AMSCs).
  Interventions: Drug: REcycled CartiLage Auto/Allo IMplantation

INTERVENTIONS:
Drug: REcycled CartiLage Auto/Allo IMplantation — Treating cartilage defects with autologous (your own) cartilage cells mixed with allogeneic (from someone else) adipose-derived mesenchymal stem cells (AMSCs).
  Other Names: RECLAIM

SUMMARY:
This is an FDA phase I study to evaluate the safety of allogeneic culture-expanded adipose-derived mesenchymal stem cells (AMSCs) combined with autologous cartilage cells to treat focal knee cartilage defects in one stage surgery.

DETAILED DESCRIPTION:
This phase I study will enroll 25 subjects with unilateral, symptomatic ICRS Grade III or IV cartilage lesions of the knee will be candidates for this study. Baseline data will include physical examination of the knee, clinical assessment of knee pain and function using validated patient reported outcome measures (PROMs), radiographs, and MRI. Tissue from qualified donors will be used to establish allogeneic MSC banks (using current Good Manufacturing Practices (cGMPs) based on standard operating procedures), which will be tested and released for clinical use. Patients will undergo surgical debridement of their cartilage defect with harvest of the articular cartilage surrounding the defect rim. Following rapid digestion into chondrocytes and their pericellular matrix, autologous chondrons will be mixed in a 1:4 ratio with allogeneic AMSCs obtained from AMSC banks and suspended in fibrin glue for application to the debrided osteochondral defect. All patients will be clinically evaluated at 1-2 weeks, 6 weeks, 12 weeks, 24 weeks, 52 weeks, 18 moths, and 24 months post-RECLAIM for adverse events (AEs). Following completion of their respective RECLAIM treatment, each subject will be followed-up for study endpoints using a predetermined protocol, including clinical evaluation, radiography, and MRI.

ELIGIBILITY:
1. Male or female ages 18-50 years.
2. Persons of childbearing potential must have a negative pregnancy test prior to receiving the study drug and will agree to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening to a period of 2 years following treatment. Females of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. A urine pregnancy test will be performed prior to the administration of the study drug to confirm negative results. If the urine pregnancy test is positive, the study drug will not be administered and the result will be confirmed by a serum pregnancy test. Urine pregnancy tests will be performed by qualified personnel using kit.
3. Persons becoming pregnant during the study will continue to be monitored for the duration of the study or completion of the pregnancy, whichever is longer. Monitoring will include perinatal and neonatal outcome. Any SAEs associated with pregnancy will be recorded.
4. Chronic (> 3 months), unilaterally symptomatic, ICRS Grade III or IV cartilage lesions ranging in size from 2 to 8 cm2. Patients with episodes of contralateral knee pain that is asymptomatic at the time of enrollment will be eligible for inclusion. However, as outlined in the primary study endpoints, patients with previous episodes of contralateral knee pain who experience a repeat episode of contralateral pain similar to their established pattern of pain during the course of the trial will not be considered as having experienced an adverse event.
5. Radiographic knee OA of Kellgren-Lawrence Grade 1 or less, consisting of normal knee radiographs (Grade 0) or doubtful narrowing of the joint space and possible osteophytic lipping (Grade 1)
6. Previous 6 week or longer trial of one of the following conservative treatments: activity modification, weight loss, physical therapy, anti-inflammatory medications or injection therapy (e.g. cortisone)
7. If applicable, at least 3 months will have passed since the last target knee intraarticular injection prior to undergoing RECLAIM therapy and at least 6 months will have passed between any prior arthroscopic or open knee procedures.
8. Able to routinely walk without assistance (e.g. cane, walker)
9. Clinically stable target knee. Patients undergoing primary anterior crucial ligament (ACL) reconstruction will be eligible for inclusion if their target knee is otherwise stable and well-aligned.
10. No additional surgery planned in the target knee for at least 12 months following RECLAIM therapy
11. Completed general physical and well-being evaluation with primary care provider within 12 months of enrollment
12. Fully understanding of the requirements of the study and willingness to comply with the treatment plan, including laboratory tests, diagnostic imaging, and follow-up visits and assessments
13. Can provide written informed consent and complete HIPAA documentation after the nature of the study is fully explained and prior to any study-related procedure 1.2 Exclusion Criteria

To be eligible for inclusion in this study, the subjects must not meet any of the following criteria:

1. Pregnant or nursing, or planning on becoming pregnant during the study period
2. Congenital or acquired malformation of the target knee resulting in significant deformity or leading to problems with the study treatment or analysis of the results
3. Significant knee malalignment that is not corrected at the time of RECLAIM surgery.
4. Injections of any kind into the target knee within 3 months prior to study enrollment
5. Greater than 50% preoperative loss in native meniscus volume (i.e. meniscectomy, degenerative loss) in the surgical knee compartment. Patients undergoing repair of meniscus tears without >50% meniscus volume loss will remain eligible for inclusion.
6. History of intra-articular infection in the target knee
7. History of superficial infection in the target knee within 6 months of study enrollment, or evidence of current superficial infection affecting the target knee
8. History of falls requiring medical attention, or gait instability
9. Clinically significant abnormal hematology (complete blood count with differential), blood chemistry, or urinalysis screening laboratory results.
10. Body mass index (BMI) > 35 kg/m2
11. Taking anticoagulant medications (e.g. warfarin, heparin or clopidogrel) which may pose a clinically-significant contraindication to surgical RECLAIM therapy
12. Taking herbal therapies or supplements within 4 weeks of enrollment or unwilling to avoid use of herbal therapies or supplements until at least 30 days following completion of the RECLAIM treatment cycle (includes, but not limited to chondroitin sulfate, diacerein, n-glucosamine, piascledine, and capsaicin)
13. Taking non-steroidal anti-inflammatory medications (e.g. COX-2 inhibitors) without a stable dosing regimen for at least 4 weeks before baseline evaluation, or anticipating not remaining on a stable dose until at least 30 days following completion of the study drug treatment cycle
14. Use of electrotherapy or acupuncture for knee pain, unless there is a stable regimen for at least 4 weeks before baseline assessment
15. Taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within 3 months prior to study enrollment
16. On chronic, immunosuppressive transplant therapy or having a chronic, immunosuppressive state, including use of systemic steroids/corticosteroids
17. Current tobacco product use, including nicotine patch or other nicotine products
18. Clinically significant systemic inflammatory, rheumatological or connective tissue disorder including but not limited to rheumatoid arthritis, systemic sclerosis, system lupus erythematosus, and Ehlers-Danlos Syndrome
19. Clinically significant rheumatological or inflammatory disease of the knee or chondrocalcinosis/calcium pyrophosphate disease (CPPD), hemochromatosis, inflammatory arthritis, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, ochronosis, hemophilic arthropath

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Nature, incidence and severity of adverse events (AEs) | 2 years
  Defined as any untoward or undesirable medical occurrence in the form of signs, symptoms, abnormal findings, or diseases that emerge or worsen relative to baseline (i.e., if present upon study entry) during the study regardless of causal relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Krych, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials